CLINICAL TRIAL: NCT07074691
Title: A Comparative Study Between Regional and Intravenous Dexamethasone in The Prophylaxis of Rebound Pain After Supraclavicular Block in Upper Limb Surgeries: A Double-Blinded Study
Brief Title: Regional and Intravenous Dexamethasone in The Prophylaxis of Rebound Pain After Supraclavicular Block in Upper Limb Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal AbdElNaby Ramadan Hamada, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS507/2/24
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Regional; Intravenous; Dexamethasone; Prophylaxis; Rebound Pain; Supraclavicular Block; Upper Limb Surgeries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional Dexamethasone group (Experimental): Patients were generally anesthetized, then a supraclavicular block is given (0.5% bupivacaine + dexamethasone 8 mg regionally), total volume = 20 mL (18 mL 0.5% bupivacaine + 2 mL dexamethasone).
  Interventions: Drug: Regional Dexamethasone
- Intravenous Dexamethasone group (Experimental): Patients were generally anesthetized, and then a supraclavicular block was administered (0.5% bupivacaine), with a total volume of 20 mL (18 mL of 0.5% bupivacaine and 2 mL of normal saline).
  Interventions: Drug: Intravenous Dexamethasone

INTERVENTIONS:
Drug: Regional Dexamethasone — Patients were generally anesthetized, then a supraclavicular block is given (0.5% bupivacaine + dexamethasone 8 mg regionally), total volume = 20 mL (18 mL 0.5% bupivacaine + 2 mL dexamethasone).
  Arms: Regional Dexamethasone group
Drug: Intravenous Dexamethasone — Patients were generally anesthetized, and then a supraclavicular block was administered (0.5% bupivacaine), with a total volume of 20 mL (18 mL of 0.5% bupivacaine and 2 mL of normal saline).
  Arms: Intravenous Dexamethasone group

SUMMARY:
This study aimed to compare the effect of regional and intravenous Dexamethasone in the prophylaxis of rebound pain after supraclavicular block in upper limb surgeries.

DETAILED DESCRIPTION:
Rebound pain is defined as "a transient acute increase in postoperative pain which occurs following resolution of a peripheral nerve block (PNB)" or as a phenomenon where a quantifiable difference is seen in the pain scores when the PNB is working compared to when its effect is resolved.

The supraclavicular block is a regional anesthetic technique used as an alternative or adjunct to general anesthesia or used for postoperative pain control for upper extremity surgeries (mid-humerus through the hand).

Dexamethasone, an adjunct used to prolong the duration of neural blockade when administered regionally or systemically, is thought to reduce pain sensitization by inhibiting sensory transmission of nociceptive C-fibers at the dorsal root ganglion and reducing prostaglandin synthesis, thereby suppressing hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) class I-II.
* Undergoing upper limb surgeries.

Exclusion Criteria:

* Patient refusal.
* History of allergy to drugs used.
* ASA class more than II ( III-IV-..).
* Uncooperative patient.
* Patients on chronic pain medications.
* Coagulopathy.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Time to the first request of analgesia | 24 hours postoperatively
  Time to the first request of analgesia was recorded from the end of surgery till the first dose of pethidine administrated.

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  All patients were familiarized with the Numeric Rating Scale (NRS) from 0 to 10, with 0 representing no pain and 10 representing maximum intolerable pain. NRS score will be assessed and recorded at 30 minutes, 2, 6, 12, 18, 24 hours postoperatively.
Patient Satisfaction | 24 hours postoperatively
  Postoperative Patient Satisfaction measured in " 4 scale patient satisfaction score" ( 1 = highly satisfied , 2 = fairly satisfied , 3 = little satisfied , 4 = non satisfied ).
Total Analgesics consumption | 24 hours postoperatively
  Pethidine 50 mg intravenous was given as postoperative rescue analgesia when the Numeric Rating Scale (NRS) score was≥ 4.
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as nausea, vomiting, hypotension and bradycardia were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.